CLINICAL TRIAL: NCT06925360
Title: The Efficacy of Intravenous Immunoglobulin for the Treatment of Bronchopulmonary Dysplasia
Brief Title: IVIG Trial for the Treatment of Bronchopulmonary Dysplasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International Peace Maternity and Child Health Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GKLW-A-2024-114-01
Record Dates: First submitted 2025-03-20; First posted 2025-04-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-11

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IVIG (Experimental)
  Interventions: Drug: intravenous immunoglobulin

INTERVENTIONS:
Drug: intravenous immunoglobulin — 1 g/kg/day for the first 2 days, 0.5 g/kg/day for next 3 days (total does 3.5 g/kg), repeatable if necessary.

SUMMARY:
It is intended to examine the efficacy and safety of intravenous immunoglobulin(IVIG) for the bronchopulmonary dysplasia in preterms. Participants will received continuous infusion IVIG 1 g/kg/day for the first 2 days, 0.5 g/kg/day for next 3 days (total does 3.5 g/kg), repeatable if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 25 weeks and 29 weeks + 6 days
* Admission within 24 hours after birth.
* Clinical symptoms and chest X-ray results show a highly suspicion of BPD.Clinical symptoms develop in several days or weeks after birth, including respiratory symptoms and signs such as shortness of breath, cyanosis or pulmonary rales, intermittent hypoxic attacks, and chronic oxygen dependence (increased oxygen concentration and assisted ventilation) .One of the following signs present in chest X-ray: lung texture thickening or ground glass opacity in early stage, diffuse lung texture blurred, lung hyperinflation, shadow of linear density increased, and shadow of triangular density increased under the pleura.
* A normal full-term newborn without a history of severe lung diseases, birth asphyxia, hypoxic-ischemic encephalopathy or other conditions that may affect the development of the respiratory, nervous and other systems.

Exclusion Criteria:

* Major congenital anomalies(e.g., congenital heart disease, congenital craniocerebral deformity, congenital structural abnormality of respiratory system, congenital hereditary metabolic disease)
* Chromosomal defects (e.g., trisomy 13, 18, 21)
* Severe intracranial hemorrhage
* Multiple organ failure
* With severe lung infections
* Other circumstances that the investigator determines are not suitable for participation in this study

Max Age: 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Survival without bronchopulmonary dysplasia at 36 weeks of postmenstrual age | 36 weeks of postmenstrual age
  For this trial, bronchopulmonary dysplasia was defined as an infant ≤32 weeks' gestational age with persistent radiographic findings of parenchymal lung disease who requires respiratory support at 36 weeks of postmenstrual age for ≥3 days to maintain arterial oxygen saturation 90%-95% .

SECONDARY OUTCOMES:
duration of mechanical ventilation | until first discharge home or 36 weeks PMA
  Defined as cumulative days on mechanical ventilation
duration of O2 supplementation | until first discharge home or 36 weeks PMA
  Defined as need for supplemental oxygen (mL/min flow or FiO2)
Time to improvement in pulmonary imaging | until first discharge home or 36 weeks PMA
Time to improvement in lung ultrasound imaging | until first discharge home or 36 weeks PMA
Preterm birth complications | until first discharge home or 36 weeks PMA
  Complications of preterm birth include retinopathy of prematurity, intraventricular hemorrhage, necrotizing enterocolitis, and septicemia et.al.
Neurodevelopmental assessment | Corrected age/ chronological age of 6 months, 1 year, and 2 years.
  Neurodevelopmental testing (e.g., Denver Developmental Screening Test)
Pulmonary function testing | Corrected age/ chronological age of 6 months, 1 year, and 2 years
  Normal/Abnormal. Pulmonary function testing includes the following parameters: Breathing Frequency (BF), Inspiratory Time (TI)/ Expiratory Time Ratio (TE), Tidal Volume (VT), Time to Peak Tidal Expiratory Flow (TPTEF), Volume to Peak Tidal Expiratory Flow (VPTEF), etc. The determination of abnormal lung function in infants is primarily relies on the analysis of TPTEF/TE and VPTEF/VE ratios, the shape of the TBFV (Tidal Breathing Flow-Volume) loop, and the integration of clinical presentation.
Vision screening | Corrected age/ chronological age of 6 months, 1 year, and 2 years
  Vision screening with Spot Vision Screener
Bone density measurement | Corrected age/ chronological age of 6 months, 1 year, and 2 years
Blood routine tests | Corrected age/ chronological age of 6 months, 1 year, and 2 years
  Including white blood cell count, differential white blood cell count (such as neutrophils, lymphocytes, etc.), red blood cell count, hemoglobin concentration, platelet count, etc
Rehabilitation evaluation | Corrected age/ chronological age of 6 months and 1 year
  e.g., Alberta Infant Motor Scale Assessment Report, 0-58 (min- max value), higher scores mean a better outcome.
Weight | Corrected age/ chronological age of 6 months, 1 year, and 2 years
Length | Corrected age/ chronological age of 6 months, 1 year, and 2 years
Head circumference | Corrected age/ chronological age of 6 months, 1 year, and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fu Xuemei, Principal Investigator — International Peace Maternity and Child Health Hospital
Locations (1):
- International Peace Maternity and Child Health Hospital, Shanghai, Shanghai Municipality, China